CLINICAL TRIAL: NCT05993026
Title: Evaluation of a School-based Intervention to Promote Mental Health and Self-efficacy Among Students in 7th to 10th Grade in Denmark: A Single-group Pre- and Post-test Design
Brief Title: A School-based Intervention to Promote Mental Health and Self-efficacy Among Students in 7th to 10th Grade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Committee for Health Education (Other); Ole Kirks Fond (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 31509
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Mental Health; Self Efficacy
Keywords: Mental Health; Self Efficacy; Schools; Students; Teachers; Teaching Materials; Denmark
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental health course (Experimental): A mental health-promoting student course offered to lower secondary school classes delivered by their teacher or another employee of the school. T
  Interventions: Behavioral: Mental health course

INTERVENTIONS:
Behavioral: Mental health course — The student course involves classroom-based teaching of eight lessons over eight weeks. The aim is to strengthen students' faith in their own abilities (self-efficacy) and ability to understand themselves and others (mentalization). In this way, students become better at entering into positive relationships and communities as well as better at handling everyday challenges both academically and socially. The student course includes teaching, exercises and training in simple tools for mastery and mentalization. The student courses in the classes are handled by staff close to the students and are based on both physical and digital material as well as an app for the students. The employees initially participate in a competency development course.

SUMMARY:
The present study is an evaluation of school-based intervention. The intervention aims to strengthen students' well-being and increase their mental health through training in tools that increase self-efficacy and ability to understand themselves and others. The Danish Committee for Health Education is responsible for developing and implementing the intervention and for recruiting schools, while the the Danish National Institute of Public Health at University of Southern Denmark is responsible for the evaluation of the intervention, including data collection, analysis and reporting.

ELIGIBILITY:
Inclusion Criteria: Student classes in grade 7 to grade 10. This corresponds to students who are typically ages between 12 and 16 years old.

Exclusion Criteria: None

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3966 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Mental wellbeing measured by the short version of the Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Measurements at baseline (one week before treatment) and follow-up (approximately 4 months after baseline)
Self-efficacy measured by two items used in the Danish Health Behaviour in School-aged Children (HBSC) study | Measurements at baseline (one week before treatment) and follow-up (approximately 4 months after baseline)
  Inspired by R. Schwarzer and M. Jerusalem two indicators to measure general self-efficacy: 'How often can you find a solution to problems if you try hard enough?' and 'How often can you manage the things you set your mind to?'

SECONDARY OUTCOMES:
Social and emotional competence | Measurements at baseline (one week before treatment) and follow-up (approximately 4 months after baseline)
  Nine items (e.g. I speak my mind when I think something is unfair), see Nielsen, L., Meilstrup, C., Nelausen, M.K., Koushede, V. and Holstein, B.E. (2015), "Promotion of social and emotional competence: Experiences from a mental health intervention applying a whole school approach", Health Education, Vol. 115 No. 3/4, pp. 339-356. https://doi.org/10.1108/HE-03-2014-0039
Student relationships | Measurements at baseline (one week before treatment) and follow-up (approximately 4 months after baseline)
  Three items from Danish Health Behaviour in School-aged Children (HBSC) study about whether the student feel (1) students in their class enjoy being together, (2) students in their class are kind and helpful and (3) accept them as they are.
Teacher support | Measurements at baseline (one week before treatment) and follow-up (approximately 4 months after baseline)
  Three HBSC items from Danish Health Behaviour in School-aged Children (HBSC) questionnaire about whether the student feel (1) accepted by their teachers, (2) that their teachers care about them as a person and (3) that they trust their teachers.
General school engagement | Measurements at baseline (one week before treatment) and follow-up (approximately 4 months after baseline)
  One HBSC item 'Liking school' from Danish Health Behaviour in School-aged Children (HBSC) questionnaire about how the student likes the school for the moment

CONTACTS AND LOCATIONS:
Overall Officials: Maj Britt Nielsen, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- The Danish Committee for Health Education, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No